CLINICAL TRIAL: NCT05023928
Title: Research on the Transformation of Postoperative Adjuvant Therapy of Tumor Antigen-sensitized DC Vaccine Applied to Esophagus Cancer
Brief Title: Tumor Antigen-sensitized DC Vaccine As an Adjuvant Therapy for Esophagus Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANT-211
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma; Esophagus Cancer
Keywords: esophagus cancer; tumor neo-antigen DC vaccine; safety; clinical efficacy
MeSH Terms: conditions — Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor antigen-sensitized DC vaccine (Experimental): Tumor antigen-sensitized vaccine is administrated, 1-week interval, totally 2 times.
  2-week later, Neo-antigen DC vaccine is administrated, 2-week interval, totally 5 times.
  Interventions: Biological: Tumor antigen-sensitized DC vaccine

INTERVENTIONS:
Biological: Tumor antigen-sensitized DC vaccine — subcutaneous administration

SUMMARY:
The aim of this single center, single arm and prospective study is to explore the safety and efficacy of tumor antigen-sensitized DC vaccine in postoperative adjuvant treatment of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of esophageal squamous cell carcinoma；
* Immunotherapy for preoperative；
* Karnofsky performance status 0-1;
* The postoperative pathological stage is (y) Pt + and / or N + M0 according to AJCC 8th
* Function of the main organs is normal;
* Edition Patient's written informed consent

Exclusion Criteria:

* Tumor emergencies;
* Abnormal coagulation function;
* Contagious diseases, such as HIV, HBV, HCV infection;
* Mental disorders;
* Concomitant tumors;
* Immunological co-morbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as events as assessed by CTCAE v4.0 | 3 months after the last administration of cells
  Number of participants with treatment-related adverse events as events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Disease-free Survival | through study completion, an average of 1 year
  Number of participants with Disease-free Survival as assessed by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu Ding, Prof, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes